CLINICAL TRIAL: NCT01021150
Title: An Open Label, Dose Escalation, Safety and Pharmacokinetics Phase 1 Study With Ombrabulin Administered as a 30-minute Intravenous Infusion in Combination With Cisplatin Administered as an Intravenous Infusion Every 3 Weeks in Patients With Advanced Solid Tumors
Brief Title: Dose Escalation, Safety and Pharmacokinetic Study of AVE8062 Combined With Cisplatin in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11088
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-06

CONDITIONS: Neoplasms, Malignant
MeSH Terms: conditions — Neoplasms | interventions — AC 7700; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ombrabulin/cisplatin (Experimental): AVE8062 combined with 75 mg/m2 of cisplatin will be administered once in every 3 weeks, with 30-minute intravenous infusion
  Interventions: Drug: ombrabulin (AVE8062); Drug: cisplatin

INTERVENTIONS:
Drug: ombrabulin (AVE8062) — Pharmaceutical form:injection solution
  Route of administration: intravenous infusion
Drug: cisplatin — Pharmaceutical form: injection solution
  Route of administration: intravenous infusion

SUMMARY:
Primary Objective:

* To determine the maximum tolerated dose based on the incidence of dose limiting toxicity and the maximum administered dose of ombrabulin in combination with cisplatin administered every 3 weeks in patients with advanced solid tumors.

Secondary Objectives:

* To assess the overall safety profile of the combination therapy.
* To characterize the pharmacokinetic profile of ombrabulin, its active metabolite RPR 258063, and cisplatin in combination.
* To evaluate anti-tumor activity of the combination therapy.

DETAILED DESCRIPTION:
The duration of the study for each patient will include an up to 4-week screening phase, 21-day study treatment cycles, an end of treatment visit and a follow-up period 30 days after the last infusion of ombrabulin. The patient will continue treatment until disease progression, unacceptable toxicity, patient's refusal of further treatment.

ELIGIBILITY:
Inclusion criteria :

* Advanced solid tumor that has become refractory to conventional treatment or for which no standard therapy exists.

Exclusion criteria :

* Eastern Cooperative Oncology Group performance status ≥ 2.
* Concurrent treatment with any other anticancer therapy
* Male or female patients who do not agree with contraception.
* Washout period of less than 28 days from prior anticancer therapies (chemotherapy, targeted agents, immunotherapy and radiotherapy) or any investigational treatment, except for nitrosoureas, mitomycin which may not be used up to 42 days prior to the first cycle.No washout period is required for hormonal therapy that has to be discontinued before the first cycle.
* Not recovered from all previous therapies (radiation, surgery, and medications). Adverse events related to previous therapies must be National Cancer Institute Common Terminology Criteria (NCI-CTCAE V3.0) grade≤1 (or alopecia≤grade 2) at screening or returned to the subject's baseline prior to their most recent previous therapy.
* Symptomatic brain metastases and carcinomatous leptomeningitis.
* Other serious illness or medical conditions not controlled by adequate treatment
* Previous cumulative carboplatin dose higher than 3,000 mg/m2 or cisplatin higher than 600 mg/m2.
* Patients whose disease has progressed or has recurred in less than 6 months from the completion of the previous platinum containing chemotherapy
* Known platinum compound hypersensitivity.
* Neuropathy and ototoxicity due to previous platinum chemotherapy.
* Inadequate organ function
* Documented medical history of myocardial infarction, documented angina pectoris, arrhythmia especially severe conduction disorder such as second or third degree atrio-ventricular block, stroke, or history of arterial or venous thrombo-embolism within the past 180 days requiring anticoagulants.
* Patient with a left ventricular ejection fraction<50% by echocardiography.
* Patients with a baseline QTc interval>0.45, or family history of Long QT Syndrome.
* Patient with uncontrolled hypertension and patient with organ damage related to hypertension such as left ventricular hypertrophy or grade 2 ocular fundscopic changes or kidney impairment.
* Patients with growing vessel disease (eg age-related macular degeneration, diabetic retinopathy, rheumatoid arthritis), or ongoing wound healing process. Patients should be enrolled in the study at least 28 days after surgery
* 12-lead Electrocardiogram: ST- and T-wave changes suggesting ischemia
* Hypertension defined as systolic blood pressure (BP)>140 mmHg or diastolic BP>90 mmHg on two repeated measurements at 30 minutes intervals.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 3 weeks (cycle 1)

SECONDARY OUTCOMES:
Global safety profile based on treatment emergent adverse events, serious adverse events, and laboratory abnormalities | on-treatment period + 30 days
Pharmacokinetic parameters of AVE8062 | Cycle 1 : Day 1 and 2; up to Cycle 4 : Day 1
Pharmacokinetic parameters of cisplatin | Day 1 to 4 of Cycle 1
Pharmacokinetic parameters of AVE8062's active metabolite RPR258063 | Cycle 1 : Day 1 and 2; up to Cycle 4 : Day 1
Objective tumor response as defined by the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | up to a maximum of 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan